CLINICAL TRIAL: NCT06682598
Title: Effects of a Multicomponent Training Based on the VIVIFRAIL Program on Functional Performance and Cognitive Function in Acutely Hospitalized Older People
Brief Title: Multicomponent Training on Functional and Cognitive Performance of Hospitalized Older People
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other); UNIVERSIDADE FEDERAL DO RIO GRANDE DO SUL (UFRGS) (Unknown)
Responsible Party: Principal Investigator, Eduardo Lusa Cadore, Associate Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: uRioGrandeHCPA
Record Dates: First submitted 2024-10-28; First posted 2024-11-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Functional Disability; Dynapenia; Cognitive Decline
Keywords: Hospitalization; Frail Older Adults; Physical Exercise; Functional Capacity
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent Training (Experimental): The subjects will perform multicomponent training sessions every day until hospital discharge day. It is composed of strength, power, balance, and walking exercises. The intervention is based on the VIVIFRAIL program, adapted for the participant's functional level.
  Interventions: Other: Multicomponent physical exercise training
- Control (No Intervention): Subjects will receive the usual care of the hospital

INTERVENTIONS:
Other: Multicomponent physical exercise training — The subjects will perform one session per day of multicomponent physical exercise training, consisting of strength, power, balance, and walking exercises. The program will have progressive intensity and volume, adapted to the frailty level of the patient. The frailty level will be screened by the Short Physical Performance Battery. Each session will consist of two strength exercises for the upper limbs and one to three for the lower limbs. Also, one exercise for balance, and walking. Participants will be instructed to perform the concentric phase of the movement as fast as possible, since a good quality of movement is maintained, and the eccentric phase in two seconds. An expert researcher will supervise the entire session.
  Arms: Multicomponent Training

SUMMARY:
The goal of this clinical trial is to determine whether a multicomponent physical exercise program improves functional and cognitive capacity in hospitalized older adults compared to the usual hospital care. The main questions it aims to answer are:

* Does a multicomponent physical exercise program improve functional and cognitive capacity?
* Is there a difference between a multicomponent physical exercise program and usual care regarding functional and cognitive outcomes after an acute hospitalization?

Researchers will compare a multicomponent physical exercise program (containing strength, balance, and walking exercises) to the usual care of the hospital to see if the program is better at maintaining or enhancing functional and cognitive outcomes

Participants will:

* Participate in multicomponent physical exercise program or receive usual care. The multicomponent group will complete the program daily for the entire hospitalization period;
* Perform functional and cognitive tests at the beginning and end of hospitalization;
* Be contacted by researchers 3, 6, and 12 months after hospital discharge.

DETAILED DESCRIPTION:
Aging is a natural and multifactorial process associated with various physiological and behavioral changes. Some of these changes can lead to increased physical inactivity, resulting in declines in functionality and increased vulnerability to diseases. During acute hospitalization, one of the several clinical consequences is excessive bedrest, even when walking is possible. Which leads to functional decline, defined as iatrogenic nosocomial disability. The literature already well describes that a multicomponent physical exercise program improves functional and cognitive capacity in frail, institutionalized, or hospitalized old people. However, a program based on this model has not yet been implemented during short-term hospitalization in Brazil. Therefore, this study aims to evaluate the effects of a multicomponent program on functional performance and cognitive function in elderly individuals with different conditions of frailty during acute hospitalization at the "Hospital de Clínicas de Porto Alegre". Functional performance will be assessed using the Short Physical Performance Battery, Timed Up and Go, 6-meter gait velocity, handgrip strength, and muscle power in 3-times-sit-to-stand. Cognitive performance will be evaluated through the Mini-Mental State Examination, Geriatric Depression Scale-15, and part "A" of the Trail Making Test. Affectiveness of the intervention will be measured using the Affectivity Scale. Participants will be randomized into two groups: multicomponent training based on VIVIFRAIL (MT) and control group. Participants in both groups will receive usual hospital treatments, including physiotherapy sessions in the morning. Participants in the MT group will perform the exercise program adjusted to their frailty and with progressive volume in the afternoon. On hospital discharge day, patients will be re-evaluated. Statistical analysis will be conducted using Generalized Estimating Equations, adopting group and time factors with two stratifications. Post-hoc LSD tests will be used to identify differences between groups. Analyses will be performed both per protocol, for individuals who complete the study, and by intention-to-treat, including those who do not complete the protocol. Results will be considered significant when p ≤ 0.05 and presented as percentage change and standard deviation with a 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or older;
* Capable of ambulating independently or with assistance;
* Pre-hospitalization Barthel Index ≥ 60;
* Does not have a terminal illness;
* Able to participate in the testing procedures and the multicomponent training program, as determined by the physician;
* Capable of providing informed consent for participation in the study.

Exclusion Criteria:

* Duration of hospitalization < 3 days;
* Lack of willingness to complete the phases of the project;
* Complications related to disease progression or intervention.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-28 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery | Baseline and immediately after the intervention
  The Short Physical Performance Battery will assess three components: static balance by having the participant stand for 10 seconds in three different positions (feet together side-by-side, semi-tandem, and tandem); gait by a 4-meter walk; and leg strength by a five-times sit-to-stand test. It ranges from zero (absence of depressive symptoms) to fifteen points (maximum score of depressive symptoms). Performance is quantified by scoring. The score ranges from 0 (functional disability) to 12 points (robust).
Timed Up and Go | Baseline and immediately after the intervention
  The Timed Up and Go test will assess dynamic balance by having the participant stand up from a chair, walk 3 meters, turn around, and return to the chair.
6-meter walk test | Baseline and immediately after the intervention
  Participants will be asked to walk a 6-meter course at their usual pace, and the time taken will be recorded.
Sit-To-Stand Muscle Power | Baseline and immediately after the intervention
  A linear encoder will assess the muscle power in the sit-to-stand test. The values of the best repetition will be considered.
Hand Grip Strength | Baseline and immediately after the intervention
  Assessed by Hand Grip Test with Hydraulic Dynamometer
Gait Symmetry | Baseline and immediately after the intervention
  Gait symmetry will be assessed by an inertial sensor. It will be obtained from the autocorrelation function of the acceleration signal along the x-axis. Gait symmetry will be considered the difference between the prominence of the first peak and the second peak after the central peak.
Gait Regularity | Baseline and immediately after the intervention
  Gait regularity will be assessed by an inertial sensor. It will be measured using the approximate entropy of the acceleration signal.
Gait Variability | Baseline and immediately after the intervention
  Gait variability will be assessed by an inertial sensor. It will be estimated by calculating the coefficient of variation of the step time.
Mini Exam of Mental State | Baseline and immediately after the intervention
  It is a screening tool used to assess cognitive function, with scoring based on a 30-point scale, where lower scores indicate greater cognitive impairment. It ranges from zero (cognitive impairment) to thirty points (good cognitive function).
Trial Making Test Part A | Baseline and immediately after the intervention
  It is an assessment of cognitive functions. In Part A, participants connect numbered circles in sequential order. The time taken to complete the task is recorded, with longer times indicating potential cognitive impairment
Geriatric Depression Scale | Baseline and immediately after the intervention
  It is a depressive symptoms scale, that consists of 15 questions with binary answers (yes/no) and is easy to understand. It ranges from zero (absence of depressive symptoms) to fifteen points (maximum score of depressive symptoms).

SECONDARY OUTCOMES:
Adherence To Intervention | Immediately after the intervention
  This will be collected by the number of sessions performed during hospitalization.
Affectivity with the intervention | Immediately after the intervention
  Will be assessed by a scale (+5 = very good, -5 = very bad).
Length of Hospitalization | Immediately after the intervention
  It will be collected through medical records
Hospital Readmission | At 3, 6, and 12 months after the intervention
  Data will be collected through telephone calls with family members at 3, 6, and 12 months following hospital discharge
Number of falls | At 3, 6, and 12 months after the intervention
  Data will be collected through telephone calls with family members at 3, 6, and 12 months following hospital discharge
Institutionalization post-hospitalization | At 3, 6, and 12 months after the intervention
  Data will be collected through telephone calls with family members at 3, 6, and 12 months following hospital discharge
Mortality | At 3, 6, and 12 months after the intervention
  Data will be collected through telephone calls with family members at 3, 6, and 12 months following hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Escola de Educação Física Fisioterapia e Dança - UFRGS, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
After the end of study, a deidentified data set will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the end of the study, no end date for sharing IPD was set.
Access Criteria: Researchers affiliated with recognized research institutions, with a research project approved by an ethics committee for the protection of human subjects, will have access to the following data: the study protocol, statistical analysis plan, informed consent form, clinical study report, and analytic code. They can request access by emailing the principal investigator with all necessary information. After review, a data table will be sent.

REFERENCES:
- [Background] Izquierdo M, Rodriguez-Manas L, Sinclair AJ. Editorial: What Is New in Exercise Regimes for Frail Older People - How Does the Erasmus Vivifrail Project Take Us Forward? J Nutr Health Aging. 2016;20(7):736-7. doi: 10.1007/s12603-016-0702-5. No abstract available. PMID 27499307
- [Background] Martinikorena I, Martinez-Ramirez A, Gomez M, Lecumberri P, Casas-Herrero A, Cadore EL, Millor N, Zambom-Ferraresi F, Idoate F, Izquierdo M. Gait Variability Related to Muscle Quality and Muscle Power Output in Frail Nonagenarian Older Adults. J Am Med Dir Assoc. 2016 Feb;17(2):162-7. doi: 10.1016/j.jamda.2015.09.015. Epub 2015 Nov 11. PMID 26577625
- [Background] Martinez-Velilla N, Casas-Herrero A, Zambom-Ferraresi F, Suarez N, Alonso-Renedo J, Contin KC, de Asteasu ML, Echeverria NF, Lazaro MG, Izquierdo M. Functional and cognitive impairment prevention through early physical activity for geriatric hospitalized patients: study protocol for a randomized controlled trial. BMC Geriatr. 2015 Sep 15;15:112. doi: 10.1186/s12877-015-0109-x. PMID 26374430
- [Background] Martinez-Velilla N, Casas-Herrero A, Zambom-Ferraresi F, Saez de Asteasu ML, Lucia A, Galbete A, Garcia-Baztan A, Alonso-Renedo J, Gonzalez-Glaria B, Gonzalo-Lazaro M, Apezteguia Iraizoz I, Gutierrez-Valencia M, Rodriguez-Manas L, Izquierdo M. Effect of Exercise Intervention on Functional Decline in Very Elderly Patients During Acute Hospitalization: A Randomized Clinical Trial. JAMA Intern Med. 2019 Jan 1;179(1):28-36. doi: 10.1001/jamainternmed.2018.4869. PMID 30419096